CLINICAL TRIAL: NCT06346704
Title: Prospective Longitudinal Monocentric Study to Evaluate the Syde® Digital Endpoint in Patients With Multiple Sclerosis (NHS-MS-EGYPT)
Brief Title: Prospective Longitudinal Monocentric Study to Evaluate the Syde® Digital Endpoint in Patients With Multiple Sclerosis
Acronym: NHS-MS-EGYPT
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision
Sponsor: SYSNAV (Industry)
Responsible Party: Sponsor
Other Study IDs: PR5030-66
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Digital Health Technology
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Digital HealthTechnology — Subject will wear the Syde® for 1 month every 6 months
  Other Names: Syde®

SUMMARY:
The study aims to assess the validity of real-world activity monitoring by the Syde® wearable device in subjects with multiple slclerosis. The Syde® collected data will be compared to on-site conventional clinical endpoints for MS pathology (EDSS, FSS and T25FWT). Subjects with multiple sclerosis will be assessed every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged from 18 to 65 years old.
2. Signed informed consent and ability to comply with study and follow-up.
3. Diagnosed with MS base on 2017 McDonald criterion
4. EDSS ≤ 5.5
5. No clinical or radiological relapse within the last 3 months
6. For patient under treatment, the molecule and its dose should be stable about 2 months before inclusion
7. Subject willing and able to comply to all study procedures including the Syde® related ones

Exclusion Criteria:

1. Patient with a cognitive or communicational disorder disturbing the understanding of the tasks or data collection
2. Previous or current disorder with an impact on current ambulation or motor function
3. Patient who have had surgery or traumatic injury in upper or lower limb within the last 6 months before the inclusion or patients who have had major surgery or trauma within the last 6 months before the inclusion

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects followed for multiple sclerosis care at the investigational site.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Longitudinal change of 95th centile of stride velocity | 2 years
  change between baseline and Month 6, Month 12, Month 18 and Month 24

SECONDARY OUTCOMES:
Correlation of the Syde® variables with the clinical assessments EDSS, FSS and T25FWT | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elnemr, MD, Principal Investigator — Air Force Specialized Hospital Cairo
Locations (1):
- Air Force Specialized Hospital, Cairo, Egypt